CLINICAL TRIAL: NCT00774852
Title: A Randomized, Double-Blind, Controlled, Phase II Multicenter Trial of CTLA4Ig (Abatacept) Plus Cyclophosphamide vs Cyclophosphamide Alone in the Treatment of Lupus Nephritis
Brief Title: Abatacept and Cyclophosphamide Combination Therapy for Lupus Nephritis
Acronym: ACCESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN034AI
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Lupus Nephritis; Lupus Erythematosus, Systemic
Keywords: lupus; systemic lupus erythematosus; lupus nephritis; SLE; abatacept; CTLA4; CTLA4Ig; glomerulonephritis
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic; Glomerulonephritis | interventions — Abatacept; Cyclophosphamide; Azathioprine; Adenosine Triphosphate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Abatacept plus Euro-lupus regimen
  Interventions: Drug: abatacept; Drug: cyclophosphamide; Drug: azathioprine; Drug: prednisone; Drug: azathioprine placebo
- Control (Placebo Comparator): Abatacept placebo plus Euro-lupus regimen
  Interventions: Drug: cyclophosphamide; Drug: azathioprine; Drug: prednisone; Drug: abatacept placebo

INTERVENTIONS:
Drug: abatacept — Intravenous infusion (500-1000 mg, dep on weight) at weeks 0, 2, and 4, then every 4 weeks until week 24; continue to week 48 only if partial response at 24 weeks
  Other Names: CTLA4Ig; Orencia
  Arms: Treatment
Drug: cyclophosphamide — 500 mg intravenous infusion every 2 weeks for 12 weeks
  Other Names: Cytoxan; Neosar
Drug: azathioprine — 2 mg/kg/day orally from weeks 12-28; continue until week 52 if only partial response observed at week 24
  Other Names: Imuran; Azasan
Drug: prednisone — 60 mg/day for 2 weeks, then taper to 10 mg/day by 12 weeks, then continue on stable dose
  Other Names: Sterapred
Drug: abatacept placebo — Intravenous infusion at weeks 0, 2, and 4, then every 4 weeks until week 24; continue to week 48 only if partial response at 24 weeks
  Arms: Control
Drug: azathioprine placebo — Oral capsule, daily from weeks 28 to 52, only if complete response observed at week 24
  Arms: Treatment

SUMMARY:
This study is for individuals with lupus who have developed complications in their kidneys, or lupus nephritis. The study will determine whether adding the experimental medication abatacept to standard cyclophosphamide therapy is more effective in improving lupus nephritis than standard cyclophosphamide therapy by itself.

DETAILED DESCRIPTION:
Lupus nephritis is an inflammation of the kidney that occurs in patients with systemic lupus erythematosus (SLE). It is caused by the immune system attacking the kidney and is among the most serious complications of SLE: left untreated it can cause long term damage to the kidneys or, in some cases, result in kidney failure.

One of the more common treatments for lupus nephritis is the "Euro-lupus" therapy. In this therapy, patients receive three different drugs - cyclophosphamide, azathioprine and prednisone - over the course of several months. However, some patients do not respond to this therapy and many only show some improvement.

In this ACCESS trial for lupus nephritis, an experimental medication known as abatacept will be added to the Euro-lupus therapy to assess if it works better than Euro-lupus therapy alone. Abatacept is a man-made protein that suppresses parts of the immune system that can cause autoimmune disease. While abatacept is experimental for lupus, it has been approved by the FDA to treat rheumatoid arthritis. Abatacept is also being studied for use in other autoimmune diseases, like multiple sclerosis and type 1 diabetes.

Participants in the ACCESS trial for lupus nephritis will receive bi-weekly intravenous infusions of cyclophosphamide for 3 months, then will take azathioprine tablets daily for at least 3 months more. Abatacept or a placebo will be administered every 2 weeks initially, then every 4 weeks for at least the first 6 months. Treatment of abatacept or placebo and azathioprine may continue for the remainder of the year. All participants will take prednisone tablets daily during the entire study.

Because the ACCESS trial is a randomized, controlled study, each participant has a 50-50 chance (like flipping a coin) of receiving abatacept. Others will receive an inactive, placebo form of the drug. Note however, that all participants will receive the Euro-lupus therapy. As a blinded (masked) study, neither participants nor study physicians will know to which group a person has been assigned.

All participants will undergo regular physical examinations, medical history and various blood and urine tests. Many of these tests will be repeated throughout the study. Participants will be asked to attend 18 study visits in the first year, and one study visit at the end of the second year.

The study will reimburse participants for certain expenses incurred as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus (SLE) by American College of Rheumatology (ACR) criteria
* Active lupus nephritis (defined by: kidney biopsy documentation within the last 12 months using International Society of Nephrology/Renal Pathology Society (ISN/RPS) classification- proliferative nephritis, active urinary sediment, urine protein-to-creatinine ratio > 1, low complement C3)
* Positive antinuclear antibody (ANA) test result at time of study entry

Exclusion Criteria:

* End stage renal disease
* Use of cyclophosphamide in the past year
* Neutropenia, thrombocytopenia, moderately severe anemia
* Active infection, including HIV, hepatitis B or C
* History of cancer, except carcinoma in situ and treated basal and squamous cell carcinomas
* Pregnant or breastfeeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wofsy, MD, Principal Investigator — University of California, San Francisco; Betty Diamond, MD, Principal Investigator — Feinstein Institute
Locations (23):
- United States (21):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Feinstein Institute, Manhasset, New York
  - Seligman Center for Advanced Therapeutics (NYU), New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Lupus Center of Excellence, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern, Dallas, Texas
- Mexico (2):
  - Unidad de investigación en enfermedades crónico - degenerativas SC, Guadalajara, Jalisco
  - El Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INNSZ), Mexico City

REFERENCES:
- [Result] ACCESS Trial Group. Treatment of lupus nephritis with abatacept: the Abatacept and Cyclophosphamide Combination Efficacy and Safety Study. Arthritis Rheumatol. 2014 Nov;66(11):3096-104. doi: 10.1002/art.38790. PMID 25403681
- [Result] Wofsy D, Diamond B, Houssiau FA. Crossing the Atlantic: the Euro-Lupus Nephritis regimen in North America. Arthritis Rheumatol. 2015 May;67(5):1144-6. doi: 10.1002/art.39067. No abstract available. PMID 25779381
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/Pages/default.aspx
- See also: Immune Tolerance Network website — http://www.immunetolerance.org
- See also: Lupus Nephritis Trials Network Research — http://lupusnephritis.org/about-the-lntn/our-research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants ages 16 and older with systemic lupus erythematosus (SLE) who met entry criteria were enrolled into the study between November 2008 and June 2012.
Groups:
- Abatacept: Subjects received abatacept IV dosed according to body weight (<60 kg, 500mg; 60-100 kg, 750 mg; or >100 kg, 1 g) at the following visits: Weeks (wks) 0, 2, and 4, then every 4 wks until Wk 24. Subjects also received: 1) cyclophosphamide 500 mg IV every 2 wks for 6 doses followed by azathioprine 2 mg/kg/day by mouth dosed by body weight at Visit 6 (rounded to the nearest 25 mg and to a maximum dose of 200 mg) for 16 wks; 2) prednisone 60 mg/day for the first 2 wks (subjects less than 60 kg could receive 1 mg/kg/day).* Prednisone was tapered until Wk 12 to a dose of 10 mg/day. This dose was continued until Wk 24 unless the subject had a prednisone-related toxicity requiring further reduction.* After Wk 24, prednisone was permitted to be tapered further to 5mg/day.* Subjects who achieved a complete response discontinued abatacept and switched to azathioprine placebo up to Wk 52 (to assess response durability). *Based on principal investigator [PI] judgment.
- Placebo: Subjects received abatacept placebo IV at the following visits: Weeks (wks) 0, 2 and 4, then every 4 wks until Wk 24. Subjects also received: 1) cyclophosphamide 500 mg IV every 2 wks for 6 doses followed by azathioprine 2 mg/kg/day by mouth dosed according to body weight at Visit 6 (rounded to the nearest 25 mg and to a maximum dose of 200 mg) for 16 wks; 2) prednisone 60 mg/day for the first two wks (subjects less than 60 kg could receive 1 mg/kg/day.*Prednisone was tapered until Wk 12 to a dose of 10 mg/day. This dose was continued until Wk 24 unless the subject had a prednisone-related toxicity that required further reduction.* After Wk 24, prednisone was permitted to be tapered further to 5mg/day.* Subjects who achieved a complete response discontinued abatacept placebo and continued azathioprine up to Wk 52. *Based on principal investigator [PI] judgment.
Period: Overall Study
Arm/Group | Abatacept | Placebo
Started | 69 | 68
Completed | 24 | 27
Not Completed | 45 | 41
Not completed — Adverse Event | 9 | 6
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 3 | 7
Not completed — Lost to Follow-up | 9 | 5
Not completed — Physician Decision | 2 | 6
Not completed — Pregnancy | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Non-responder | 15 | 11
Not completed — Subject non-compliance | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Subject received prohibited medication | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat sample
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 65 | 67 | 132
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (10.1) | 32.7 (12.0) | 32.4 (11.1)
Age, Customized [Number; unit: participants]
  <18 Years | 1 | 0 | 1
  18-20 Years | 7 | 5 | 12
  21-24 Years | 10 | 15 | 25
  >24 Years | 48 | 48 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 64 | 122
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 58 | 59 | 117
  Mexico | 8 | 9 | 17
Duration of Lupus Nephritis [Number; unit: participants] — Years since lupus nephritis was diagnosed by a physician. This information was obtained by medical history during the Baseline Visit.
  participants
    <1 Year | 47 | 48 | 95
    >=1 Year | 19 | 20 | 39
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] — The highest serum creatinine reading from either screening or baseline visit was used for this measure. According to Harrison's Principles of Internal Medicine, normal results are 0.6 to 1.2 mg/dL for men and 0.5 to 0.9 mg/dL for women. This test measures kidney function. Abnormal kidney function results in increased levels of serum creatinine.
  mg/dL | 1.3 (0.7) | 1.2 (0.6) | 1.2 (0.7)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Estimated glomerular filtration rate (eGFR) is a calculation based on serum creatinine result, age, sex and race. GFR is a marker of kidney function. Normal GFR is approximately 100mL/min/1.73m^2. Lower GFRs reflect poorer kidney function.
  mL/min/1.73m^2 | 64.6 (36.2) | 58.4 (27.8) | 61.4 (32.2)
Urine Protein (24 hour collection) [Mean (Standard Deviation); unit: mg/day] — Several measures of kidney (renal) function were obtained from a 24 hour urine collection: urine protein (mg/day), -creatinine (mg/day), -protein: -creatinine ratio (mg:mg). Urine protein normal values: less than 80 mg/day. Greater levels of urine protein may indicate kidney disease.
  mg/day | 3814.8 (3063.6) | 4509.4 (3987.7) | 4167.3 (3566.4)
Urine Creatinine (24 hour collection) [Mean (Standard Deviation); unit: mg/day] — Several measures of kidney (renal) function were obtained from a 24 hour urine collection: urine protein (mg/day), -creatinine (mg/day), -protein: -creatinine ratio (mg:mg). Urine creatinine normal range: 500 to 2000 mg/day. An abnormal result may indicate poorer kidney function.
  mg/day | 1081.5 (532.4) | 1132.8 (409.3) | 1107.6 (472.8)
Urine Protein-to-Creatinine Ratio (24 hour collection) [Mean (Standard Deviation); unit: mg:mg] — Several measures of kidney (renal) function were obtained from a 24 hour urine collection: urine protein (mg/day), -creatinine (mg/day), -protein: -creatinine ratio (mg:mg). Urine protein-to-creatinine ratio is an indicator of proteinuria. A ratio greater than 0.2 mg:mg is considered an indicator of poor kidney function.
  mg:mg | 3.6 (2.6) | 4.1 (3.4) | 3.9 (3.0)
Urine Protein-to-Creatinine Ratio [Number; unit: participants] — Urine protein: creatinine ratio is a comparison of protein to creatinine in urine which is an indicator of proteinuria. A ratio greater than 0.2 mg:mg is considered an indicator of poor kidney function. Participants are stratified as either 1.) greater than or 2.) <=3 mg:mg.
  participants
    > 3 mg:mg | 27 | 31 | 58
    <= 3 mg:mg | 39 | 37 | 76
Average Daily Prednisone Dose [Mean (Standard Deviation); unit: mg/day] — Average daily prednisone dose taken by participants during 14 days prior to initiation of study drug.
  mg/day | 47.0 (18.5) | 39.0 (20.3) | 42.8 (19.8)
Anti-dsDNA [Number; unit: participants] — Participants with systemic lupus erythematosus (SLE) may have autoantibodies (e.g., self against self) to double-stranded DNA. Double-stranded DNA is one of multiple diagnostic tests for SLE and levels may be associated with disease activity. A positive test for autoantibodies to double-stranded DNA is based on the normal range from the local laboratory. Baseline is defined as the last measurement taken on or prior to the first day of dosing. Not all subjects had available data.
  participants
    Negative | 14 | 15 | 29
    Equivocal ("borderline") | 2 | 2 | 4
    Positive | 49 | 50 | 99
Serum Complement Test C3 [Mean (Standard Deviation); unit: mg/dL] — Serum complement tests (complement C3, -C4 and -CD50) measure a group of proteins in the blood. Low blood levels of complement are common in people who have active lupus. Harrison's Principles of Internal Medicine normal values: C3 83 - 177 mg/dL.
  mg/dL | 64.2 (25.5) | 70.4 (30.4) | 67.3 (28.1)
Serum Complement Test C4 [Mean (Standard Deviation); unit: mg/dL] — Serum complement tests (complement C3, -C4 and -CD50) measure a group of proteins in the blood. Low blood levels of complement are common in people who have active lupus. Harrison's Principles of Internal Medicine normal values: C4 = 16 - 47 mg/dL.
  mg/dL | 13.0 (8.9) | 13.4 (6.8) | 13.2 (7.9)
Serum Complement Test CH50 [Mean (Standard Deviation); unit: units/mL] — Serum complement tests (complement C3, -C4 and -CD50) measure a group of proteins in the blood. Low blood levels of complement are common in people who have active lupus. Harrison's Principles of Internal Medicine normal values: CD50 (a measure of total complement activity) 41 - 90 hemolytic units/mL.
  units/mL | 47.0 (41.3) | 61.3 (52.2) | 54.3 (47.5)
Participants with Hypocomplementemia [Number; unit: participants] — Participants were categorized as having hypocomplementemia if their serum complement test results (C3, C4 and/or CH50) were below the normal range at the site. Below normal complement test results are indicative of active lupus erythematosus.Not all subjects had available data.
  participants
    C3 hypocomplementemia | 47 | 44 | 91
    C4 hypocomplementemia | 39 | 37 | 76
    CH50 hypocomplementemia | 29 | 23 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Complete response definition: a serum creatinine <= 1.2 mg/dL or <=125% of the higher value at either screening or baseline visit, protein-to-creatinine ratio <0.5, and prednisone dose tapered to <=10 mg/day or prednisone dosing allowances in protocol. Participants had to meet all of the referenced criteria to be considered a complete responder (CR). Participants who discontinued treatment and/or terminated from the study in the first 24 weeks were defined as CR failures for all subsequent visits. CRs are those who successfully responded to treatment and have minimal activity of their lupus nephritis.
Time Frame: Week 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 66 | 68
participants | 22 | 21
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority or Other; p = 0.85, Chi-squared; Two-sided Pearson's chi-square test

2. Secondary Outcome: Number of Participants With Partial Response
Description: Outcome measure description: Partial response definition: a serum creatinine <= 1.2 mg/dL or <= to 125% of the higher value at either screening or baseline visit, and improvement (reduction) >= to 50% in the urine protein to creatinine ratio at either screening or baseline visit, and prednisone dose has been tapered to 10 mg/day or according to protocol dosing allowances in protocol. Participants who discontinued treatment and/or terminated from the study in the first 24 weeks were defined as complete response failures for all subsequent visits. Partial responders are those who showed some response to treatment and low activity of their lupus nephritis.
Time Frame: Week 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 66 | 68
participants | 39 | 40
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority or Other; p = 0.99, Chi-squared; Two-sided Pearson's chi-square test

3. Secondary Outcome: Number of Participants With a Complete or Partial Response
Description: Complete response: a serum creatinine <= 1.2 mg/dL or <=125% of the higher value at either screening or baseline visit, protein-to-creatinine ratio <0.5, and prednisone dose tapered to <=10 mg/day or prednisone dosing allowances in protocol. Participants had to meet all of the referenced criteria to be considered a complete responder.
  Partial response: a serum creatinine <= 1.2 mg/dL or <= to 125% of the higher value at either screening or baseline visit, and improvement >= to 50% in the urine protein to creatinine ratio at either screening or baseline visit, and prednisone dose has been tapered to 10 mg/day or according to protocol dosing allowances in protocol.
  Participants who discontinued treatment and/or terminated from the study were defined as response failures for all subsequent visits. CRs successfully responded to treatment and have minimal activity of their lupus nephritis. Partial responders showed some response to treatment and low activity of their lupus nephritis.
Time Frame: Week 52
Population: Intent-to-treat
Measure: Number; unit: participants
Groups:
- Week 24 Complete Response: Abatacept: At Week 28 participants assigned to Abatacept group who were classified as a complete responder at their Week 24 visit discontinued abatacept and switched to overencapsulated azathioprine placebo up to Week 52
- Week 24 Complete Response: Placebo: At Week 28 participants assigned to the Placebo group who were classified as a complete responder at their Week 24 visit discontinued abatacept placebo and switched to overencapsulated azathioprine up to Week 52
- Week 24 Partial Response: Abatacept: At Week 28 participants assigned to Abatacept group who were classified as a partial responder at their Week 24 visit continued to receive abatacept up to Week 48 and azathioprine up to Week 52
- Week 24 Partial Response: Placebo: At Week 28 participants assigned to the Placebo group who were classified as a partial responder at their Week 24 visit continued to receive abatacept placebo up to Week 48 and azathioprine up to Week 52
Arm/Group | Week 24 Complete Response: Abatacept | Week 24 Complete Response: Placebo | Week 24 Partial Response: Abatacept | Week 24 Partial Response: Placebo
Number analyzed (Participants) | 22 | 21 | 17 | 19
participants | 12 | 14 | 13 | 13
Statistical Analysis 1: Comparison: Week 24 Complete Response: Abatacept vs Week 24 Complete Response: Placebo; Test type: Superiority or Other; p = 0.54, Chi-squared; Two-sided Pearson's chi-square test
Statistical Analysis 2: Comparison: Week 24 Partial Response: Abatacept vs Week 24 Partial Response: Placebo; Test type: Superiority or Other; p = 0.72, Chi-squared; Two-sided Pearson's chi-square test

4. Secondary Outcome: Number of Participants Who Achieved a Complete Response by Week 24 and Maintained the Complete Response Through Week 52
Description: Complete response definition: a serum creatinine <= 1.2 mg/dL or <=125% of the higher value at either screening or baseline visit, protein-to-creatinine ratio <0.5, and prednisone dose tapered to <=10 mg/day or prednisone dosing allowances in protocol. Participants had to meet all of the referenced criteria to be considered a complete responder (CR). Participants who discontinued treatment and/or terminated from the study were defined as response failures for all subsequent visits. CRs are those who successfully responded to treatment and had minimal activity of their lupus nephritis.
Time Frame: Week 52
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Week 24 Complete Response: Abatacept | Week 24 Complete Response: Placebo
Number analyzed (Participants) | 22 | 21
participants | 11 | 13
Statistical Analysis 1: Comparison: Week 24 Complete Response: Abatacept vs Week 24 Complete Response: Placebo; Test type: Superiority or Other; p = 0.54, Chi-squared; Two-sided Pearson's chi-square test

5. Secondary Outcome: Number of Participants Fulfilling the Proteinuria and Prednisone Criteria of a Complete Response
Description: A complete proteinuria and prednisone response is defined as urine protein-to-creatinine ratio <0.5 and prednisone dose tapered to <= 10mg/day. Subjects who discontinued treatment or terminated from the study in the first 24 weeks are defined as response failures for all subsequent visits. Complete responders are those who successfully responded to treatment and have minimal activity of their lupus nephritis.
Time Frame: Week 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 66 | 68
participants | 22 | 21

6. Secondary Outcome: Number of Participants Fulfilling the Proteinuria and Prednisone Criteria of a Partial Response
Description: A partial proteinuria and prednisone response is defined as an improvement (reduction) of >=50% in the urine protein-to-creatinine ratio at either visit -1 or 0, and prednisone dose has been tapered to 10 mg/day. Subjects who discontinued treatment or terminated from the study in the first 24 weeks are defined as response failures for all subsequent visits. Partial responders are those who showed some response to treatment and low activity of their lupus nephritis.
Time Frame: Week 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 66 | 68
participants | 39 | 42

7. Secondary Outcome: Number of Participants Who Achieved No Response at 24 Weeks and Continued in the Study
Description: A participant who did not meet the criteria for either a complete response or a partial response at Week 24 was considered a non-responder. After Week 24, non-responders were terminated from the study and treated according to best clinical judgment unless the site investigator judged that the participant could benefit from continued participation. Non responders did not respond to treatment and lupus activity is moderate to severe.
Time Frame: Week 104
Population: Intent-to-treat
Measure: Number; unit: participants
Groups:
- Week 24 Non-Responder: Abatacept: Participants who were in the abatacept arm and non-responders at Week 24 either terminated or continued participation. If participation continued, participants continued abatacept up to Week 48 and azathioprine up to Week 52
- Week 24 Non-Responder: Placebo: Participants who were in the placebo arm and non-responders at Week 24 either terminated or continued participation. If participation continued, participants continued abatacept placebo up to Week 48 and azathioprine up to Week 52
Arm/Group | Week 24 Non-Responder: Abatacept | Week 24 Non-Responder: Placebo
Number analyzed (Participants) | 15 | 11
participants | 0 | 0

8. Secondary Outcome: Number of Participants Who Achieved No Response at 24 Weeks and Continued in the Study , Achieving a Complete or Partial Response
Description: A participant who did not meet the criteria for either a complete response (CR) or a partial response (PR) at Week 24 was considered a non-responder. After Week 24, non-responders were terminated from the study and treated according to best clinical judgment unless the investigator judged that the participant may benefit from continued participation. CR definition: a serum creatinine <= 1.2 mg/dL or <=125% of the higher value at either screening or baseline visit, protein-to-creatinine ratio <0.5, and prednisone dose tapered to <=10 mg/day or prednisone dosing allowances in protocol. Participants had to meet all of the referenced criteria to be considered a CR. PR definition: a serum creatinine <= 1.2 mg/dL or <= to 125% of the higher value at either screening or baseline, and improvement (reduction) >= to 50% in the urine protein to creatinine ratio at either screening or baseline, and prednisone dose has been tapered to 10 mg/day.
Time Frame: Week 52
Population: Intent-to-treat
Groups:
- Week 24 Non-Responder Who Continued Treatment: Abatacept: Participants who were in the abatacept arm and non-responders at Week 24 who continued participation. If participation continued, participants continued abatacept up to Week 48 and azathioprine up to Week 52
- Week 24 Non-Responder Who Continued Treatment: Placebo: Participants who were in the placebo arm and non-responders at Week 24 who continued participation. If participation continued, participants continued abatacept placebo up to Week 48 and azathioprine up to Week 52
Arm/Group | Week 24 Non-Responder Who Continued Treatment: Abatacept | Week 24 Non-Responder Who Continued Treatment: Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Lupus Disease Activity - Participants Who Were Anti-dsDNA Positive at Baseline and Negative at Week 104
Description: Lupus disease activity was assessed by 7 different measures: reduction in anti-dsDNA, negative anti-dsDNA, resolution of hypocomplementemia (C3, C4), frequency of flares, patient global assessment, SF36 total scores, and BILAG-2004 scores.
  Participants with systemic lupus erythematosus (SLE) may have autoantibodies (e.g., self against self) to double-stranded DNA. Double-stranded DNA is one of multiple diagnostic tests for SLE and levels may be associated with disease activity. One measure used to assess disease activity is the number of participants who were anti-dsDNA positive at baseline but negative at Week 104. Going from positive to negative is indicative of lowered lupus activity.
Time Frame: Week 104
Population: Participants from Intent-to-treat population who had positive anti-dsDNA at baseline and completed Week 104.
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 18 | 18
participants | 3 | 3
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Comparison of Participants across groups who had negative anti-dsDNA at Week 104. Baseline is defined as the last measurement taken on or prior to the first day of dosing. Analysis is performed on participants with available data; Test type: Superiority or Other; p > 0.99, Chi-squared; Two-sided Pearson's chi-squared test

10. Secondary Outcome: Lupus Disease Activity - Negative Anti-dsDNA
Description: Lupus disease activity was assessed by 7 different measures: reduction in anti-dsDNA, negative anti-dsDNA, resolution of hypocomplementemia (C3, C4), frequency of flares, patient global assessment, SF36 total scores, and BILAG-2004 scores.
  Participants with systemic lupus erythematosus (SLE) may have autoantibodies (e.g., self against self) to double-stranded DNA. Double-stranded DNA is one of multiple diagnostic tests for SLE and levels may be associated with disease activity. This measure was the number of participants who had negative anti-dsDNA at Week 104. Having a negative score is indicative of low lupus disease activity.
Time Frame: Week 104
Population: Intent-to-treat participants who completed Week 104.
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 24 | 27
participants | 7 | 10
Statistical Analysis 1: Comparison: Abatacept vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p > 0.99, Chi-squared; Two-sided Pearson's chi-squared test

11. Secondary Outcome: Lupus Disease Activity - Presence of Hypocomplementemia
Description: Lupus disease activity was assessed by 7 different measures: anti-dsDNA, negative anti-dsDNA, resolution of hypocomplementemia (C3, C4), frequency of flares, patient global assessment, SF36 total scores, and BILAG-2004 scores.
  Participants were categorized as having hypocomplementemia if their serum complement test results (C3, and C4) were below the normal range at the site. Below normal complement test results are indicative of active lupus erythematosus.
Time Frame: Week 104
Population: Intent-to-treat participants who completed Week 104 and had hypocomplementemia data available
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 23 | 27
participants
  C3 Hypocomplementemia | 12 | 11
  C4 Hypocomplementemia | 11 | 8

12. Secondary Outcome: Lupus Disease Activity - Frequency of Flares
Description: Lupus disease activity was assessed by 7 different measures: anti-dsDNA, negative anti-dsDNA, resolution of hypocomplementemia (C3, C4), frequency of flares, patient global assessment, SF36 total scores, and BILAG-2004 scores.
  Flares can be renal or non-renal. A renal flare is defined as two successive evaluations at least 1 week apart as proteinuria >1 gm/24h for participants who attain a complete response at Week 12 and for all other participants either 1) Increasing serum creatinine and persistent proteinuria, or 2) Worsening proteinuria. A non-renal flare is defined as any new post-baseline BILAG A in a non-renal organ system using BILAG-2004. This outcome measures the number of participants with the presence of renal and non-renal flares from Week 24 through Week 52 by response status. Having flares is indicative of more lupus disease activity.
Time Frame: Week 52
Population: Intent-to-treat with available data between weeks 24 and 52.
Measure: Number; unit: participants
Groups:
- Week 24 No Response: Abatacept: At Week 28 participants assigned to Abatacept group who were classified as a non-responder at their Week 24 visit either terminated from the study at Wk 28 or continued to receive abatacept up to Week 48 and azathioprine up to Week 52, at the discretion of the investigators
- Week 24 No Response: Placebo: At Week 28 participants assigned to Placebo group who were classified as a non-responder at their Week 24 visit either terminated from the study at Wk 28 or continued to receive abatacept placebo up to Week 48 and azathioprine up to Week 52, at the discretion of the investigators
Arm/Group | Week 24 Complete Response: Abatacept | Week 24 Complete Response: Placebo | Week 24 Partial Response: Abatacept | Week 24 Partial Response: Placebo | Week 24 No Response: Abatacept | Week 24 No Response: Placebo
Number analyzed (Participants) | 22 | 21 | 17 | 19 | 14 | 11
participants
  Participants with a Renal Flare | 0 | 2 | 1 | 3 | 1 | 0
  Participants with at least 1 Non-renal Flare | 1 | 1 | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Week 24 Complete Response: Abatacept vs Week 24 Complete Response: Placebo; Comparison of groups with renal flare; Test type: Superiority or Other; p = 0.23, Chi-squared; Pearson's
Statistical Analysis 2: Comparison: Week 24 Partial Response: Abatacept vs Week 24 Partial Response: Placebo; Comparison of groups with renal flare; Test type: Superiority or Other; p = 0.61, Chi-squared; Pearson's
Statistical Analysis 3: Comparison: Week 24 Complete Response: Abatacept vs Week 24 Complete Response: Placebo; Comparison of groups with at least one non-renal flare; Test type: Superiority or Other; p > 0.99, Chi-squared; Pearson's
Statistical Analysis 4: Comparison: Week 24 Partial Response: Abatacept vs Week 24 Partial Response: Placebo; Comparison of groups with at least one non-renal flare; Test type: Superiority or Other; p > 0.99, Chi-squared; Pearson's

13. Secondary Outcome: Lupus Disease Activity - Patient Global Assessment
Description: Lupus disease activity was assessed by 7 different measures: anti-dsDNA, negative anti-dsDNA, resolution of hypocomplementemia (C3, C4), frequency of flares, patient global assessment (PGA), SF36 total scores, and BILAG-2004 scores.
  PGA is measured on a 100mm scale and assessed at Weeks 0, 12, 24, 52, and 104. Higher values indicate greater burden of disease.
Time Frame: Week 104
Population: Intent-to-treat who completed Week 104 and had patient global assessment data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 24 | 26
units on a scale | 13.2 (19.5) | 18.7 (26.7)

14. Secondary Outcome: Lupus Disease Activity - Patient Global Assessment Percent Change From Baseline
Description: as for outcome 13
Time Frame: Week 104
Population: Intent-to-treat who completed Week 104 and had patient global assessment data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 24 | 26
percent change | 26 (343.9) | -35.2 (98.0)

15. Secondary Outcome: Lupus Disease Activity - SF-36 Scores
Description: Lupus disease activity was assessed by 7 different measures: anti-dsDNA, negative anti-dsDNA, resolution of hypocomplementemia (C3, C4), frequency of flares, patient global assessment, SF36 total scores, and BILAG-2004 scores.
  The SF-36 is a quality of life assessment that was performed at Weeks 9, 24, 36, 52, and 104. Eight scale scores are derived from responses to the 36 items of the SF-36 questionnaire which were combined to produce the Physical Component Score and the Mental Component Score. The Physical Component Score is based on the Physical Functioning Scale (10 items), the Role-Physical Scale (4 items), the Bodily Pain Scale (2 items), and the General Health Scale (5 items). The Mental Component Score is based upon the Vitality Scale (4 items), the Social Functioning Scale (2 items), the Role-Emotional Scale (3 items) and the Mental Health Scale (5 items). Each component score is transformed into a 0-100 scale, with higher numbers indicating greater quality of life.
Time Frame: Week 104
Population: Intent-to-treat who completed Week 104 and had SF-36 data available.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 24 | 27
Score
  Week 104 Physical Component Score | 49.3 (11.1) | 45.3 (11.8)
  Week 104 Mental Component Score | 50.9 (12.7) | 49.2 (12.4)

16. Secondary Outcome: Lupus Disease Activity - SF-36 Scores Percent Change From Baseline
Description: as for outcome 15
Time Frame: Week 104
Population: Intent-to-treat who completed Week 104 and had SF-36 data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 24 | 26
percent change
  Percent Change From Baseline on Physical Component | 32.1 (49.1) | 28.2 (66.4)
  Percent Change from Baseline Mental Component Scor | 39.6 (70.4) | 37.1 (55.2)

17. Secondary Outcome: Lupus Disease Activity - Total BILAG-2004
Description: BILAG-2004 has 5 categories of scoring.Category A:defined by severe disease activity requiring any of the following treatments: 1) systemic high dose oral glucocorticoids, 2) IV pulse glucocorticoids, 3) systemic immunomodulators, or 4)therapeutic high dose anticoagulation in the presence of high dose steroids or immunomodulators. Category B:defined by moderate disease activity requiring any of the following treatments:1) systemic low dose oral glucocorticoids, 2) intramuscular or intra-articular or soft tissue glucocorticoids injection,3) topical glucocorticoids, 4) topical immunomodulators,5) antimalarials or thalidomide or prasterone or acitretin, or 6) symptomatic therapy.Category C:defined by mild disease.Category D is defined by inactive disease, previously affected.Category E is defined as the system never being involved.The categories are converted to a numeric score (A=9, B=3, C=1, D=0, E=0) and treated as a continuous variable. Higher score= more severe disease activity.
Time Frame: Week 52
Population: Intent-to-treat who completed Week 52 and BILAG 2004 data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 24 Complete Response: Abatacept | Week 24 Complete Response: Placebo | Week 24 Partial Response: Abatacept | Week 24 Partial Response: Placebo
Number analyzed (Participants) | 14 | 16 | 14 | 14
units on a scale | 1.8 (1.4) | 1.9 (1.6) | 3.2 (2.6) | 3.5 (1.8)
Statistical Analysis 1: Comparison: Week 24 Complete Response: Abatacept vs Week 24 Complete Response: Placebo; Test type: Superiority or Other; p = 0.79, ANCOVA — P-value compares actual values between experimental and control groups at Week 52 and is derived from two-sided t-test from and ANCOVA model that adjusts for baseline values
Statistical Analysis 2: Comparison: Week 24 Partial Response: Abatacept vs Week 24 Partial Response: Placebo; Test type: Superiority or Other; p = 0.74, ANCOVA — [p-value comment as in outcome 17, analysis 1]

18. Secondary Outcome: Proportion of Vaccinated Participants With a Competent Immune Response
Description: Among participants who are vaccinated, the number of who have a competent immune response at Week 52 as defined as having met both of the following criteria:
  1. Pneumococcal vaccination response - absolute value >= 0.35 ug/mL and, when measured 4-6 weeks after vaccination, a >=2-fold increase from baseline in serotype-specific antibody titer for at least 50% of the serotypes tested.
  2. Tetanus toxoid vaccination response - absolute value >=0.015 IU/mL and, when measured 4-6 weeks after vaccination, a 2-fold increase from baseline in antigen-specific antibody titer
  Competent immune response is indicative of low disease activity.
Time Frame: Week 52
Population: Intent-to-treat who completed Week 52 and were vaccinated.
Measure: Number; unit: percentage of participants
Arm/Group | Week 24 Complete Response: Abatacept | Week 24 Complete Response: Placebo
Number analyzed (Participants) | 3 | 4
percentage of participants
  Pneumococcal Vaccines | 67 | 100
  Tetanus Toxoid Vaccines | 50 | 100
Statistical Analysis 1: Comparison: Week 24 Complete Response: Abatacept vs Week 24 Complete Response: Placebo; Comparison of groups for Pneumococcal vaccines; Test type: Superiority or Other; p = 0.43, Chi-squared; Pearson's
Statistical Analysis 2: Comparison: Week 24 Complete Response: Abatacept vs Week 24 Complete Response: Placebo; Comparison of groups for Tetanus Toxoid vaccines; Test type: Superiority or Other; p = 0.99, Chi-squared; Pearson's

ADVERSE EVENTS:
Time Frame: From enrollment through last follow-up visit (up to 104 weeks)
Arm/Group | Abatacept | Placebo
Serious Adverse Events (participants affected / at risk) | 28/69 | 26/68
Other Adverse Events (participants affected / at risk) | 39/69 | 42/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=69) | Placebo (N=68)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Lupus myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral myocarditis (Infections and infestations) | 0 (0) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (5)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hemisensory neglect (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=69) | Placebo (N=68)
Leukopenia (Blood and lymphatic system disorders) | 10 (13) | 8 (9)
Nausea (Gastrointestinal disorders) | 7 (8) | 6 (13)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3)
Adverse drug reaction (General disorders) | 3 (3) | 5 (6)
Oedema peripheral (General disorders) | 6 (6) | 3 (3)
Bronchitis (Infections and infestations) | 5 (5) | 3 (4)
Herpes zoster (Infections and infestations) | 4 (4) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 12 (17)
Urinary tract infection (Infections and infestations) | 4 (7) | 9 (11)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Chest pain (General disorders) | 0 (0) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No